CLINICAL TRIAL: NCT02403505
Title: Conducting an Early Phase Clinical Trial to Assess for CEA Antigen Presentation Therapeutic Biological Product Mix Activity That Suggests the Potential for Clinical Benefits of CEA Positive Rectal Cancer Patients.
Brief Title: Early Phase Clinical Trial About Therapeutic Biological Product Mix for Treating CEA Positive Rectal Cancer
Acronym: CEA+RC-BCG
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Han Xu, M.D., Ph.D., FAPCR, Sponsor-Investigator, IRB Chair (Industry)
Collaborators: UnitedHealthcare (Other)
Responsible Party: Sponsor-Investigator, Han Xu, M.D., Ph.D., FAPCR, Sponsor-Investigator, IRB Chair, M.D., Ph.D., FAPCR, Sponsor-Investigator, Medical Director, IORG Director, Medical Monitor, Safety Officer, IRB Chair, Medicine Invention Design, Inc
Organization: Medicine Invention Design, Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IND 009549; FWA00015357 (Registry Identifier: HHS, Human Protections Administrator); IORG0007849 (Registry Identifier: HHS, IORG); IRB00009424 (Registry Identifier: HHS, IRB); NPI-1831468511 (Registry Identifier: HHS, Health Care Provider Individual); NPI-1023387701 (Registry Identifier: HHS, Health Care Provider Organization); IND 009549 (Registry Identifier: FDA, Investigational New Drug Application (IND))
Record Dates: First submitted 2015-03-15; First posted 2015-03-31 (Estimated); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Rectal Cancer
Keywords: CEA; Antigen Presentation; APC; Trained Immunity; Innate Immune Memory; Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: * Single Usage
  * Single Dosage
Masking Description: Open Label
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Assess for CEA Antigen Presentation Therapeutic Biological Product Mix activity (Experimental): CEA protein antigen 0.05 mg add into BCG Organism 50 MG
  Interventions: Biological: CEA protein antigen plus BCG Vaccine Mix for percutaneous use

INTERVENTIONS:
Biological: CEA protein antigen plus BCG Vaccine Mix for percutaneous use — * By the percutaneous route with the multiple puncture device
  * CEA protein antigen 0.05 mg plus BCG Organism 50 MG Mix
  Other Names: CEA protein antigen plus BCG Organism Mix

SUMMARY:
Conducting an early phase clinical trial to assess CEA Antigen Presentation Therapeutic Biological Product Mix activity that suggests the potential for clinical benefit of CEA positive rectal cancer patients.

1. Treat CEA positive rectal cancer via Trained Immunity.
2. Activate human CEA Protein Antigen Presentation Reaction.
3. The human antigen presenting cells (APCs) can treat the CEA protein antigen into small peptide fragments, and then kill CEA positive rectal cancer cells in vivo.

DETAILED DESCRIPTION:
* Conducting an early phase clinical trial to assess CEA Antigen Presentation Therapeutic Biological Product Mix activity that suggests the potential for clinical benefit of CEA positive rectal cancer patients
* 20 CEA Positive Rectal Cancer Patients
* Positive testing CEA by blood-drawing
* TB negative participant is negative IGRA blood test with TB antigens
* Clinical Rectal Cancer Diagnosis Stage 0 - IIA
* Clinical Rectal Cancer Diagnosis without symptoms
* Clinical Rectal Cancer Diagnosis without metastasis
* CEA protein antigen 0.05 mg plus BCG Organism 50 MG Mix
* By the percutaneous route with the multiple puncture device
* Positive IGRA blood test with CEA protein antigen after percutaneous use 21 days
* Our trial duration will be 12-week duration

ELIGIBILITY:
Conducting an early phase clinical trial to assess CEA Antigen Presentation Therapeutic Biological Product Mix that suggests the potential for clinical benefit of CEA positive rectal cancer patients.

20 CEA Positive Rectal Cancer Patients

Inclusion Criteria:

* Clinical Rectal Cancer Diagnosis Stage 0 - IIA
* Clinical Rectal Cancer Diagnosis without symptoms
* Clinical Rectal Cancer Diagnosis without metastasis
* Positive testing CEA by blood-drawing
* TB negative participant is negative IGRA blood test with TB antigens.

Exclusion Criteria:

* Pregnant
* Thrombosis
* Allergy
* TB positive participant is positive IGRA blood test with TB antigens.
* Symptoms of rectal cancer
* Metastasis of rectal cancer
* Evidence of critical illness

Ages: 24 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-12-28 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
20 Rectal Cancer Participants with CEA blood test | Duration up to 90 days
  Positive testing CEA by blood-drawing
20 Rectal Cancer Participants with IGRA blood test with CEA protein antigen | Duration up to 90 days
  Positive IGRA blood test with CEA protein antigen after percutaneous use 21 days
20 Rectal Cancer Participants with IGRA blood test with TB antigens | Duration up to 90 days
  * Negative IGRA blood test with TB antigens before percutaneous use
  * Positive IGRA blood test with TB antigens after percutaneous use 21 days

CONTACTS AND LOCATIONS:
Overall Officials: HAN XU, MD/PhD/FAPCR, Study Chair — IRB00009424--NPI-1831468511; HAN XU, MD/PhD/FAPCR, Study Director — IORG0007849--NPI-1023387701; HAN XU, MD/PhD/FAPCR, Principal Investigator — IORG0007849--FWA00015357
Locations (1):
- Medicine Invention Design, Inc. (MIDI) - c/o - IORG0007849 - NPI-1023387701, Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: IORG0007849 — http://ohrp.cit.nih.gov/search/search.aspx?styp=bsc
- See also: IRB00009424 — http://ohrp.cit.nih.gov/search/search.aspx?styp=bsc
- See also: FWA00015357 — http://ohrp.cit.nih.gov/search/search.aspx?styp=bsc

DOCUMENTS (3):
  • Study Protocol (2024-08-27): https://cdn.clinicaltrials.gov/large-docs/05/NCT02403505/Prot_014.pdf
  • Statistical Analysis Plan (2024-08-27): https://cdn.clinicaltrials.gov/large-docs/05/NCT02403505/SAP_015.pdf
  • Informed Consent Form (2024-08-27): https://cdn.clinicaltrials.gov/large-docs/05/NCT02403505/ICF_016.pdf